CLINICAL TRIAL: NCT00739752
Title: Interventions to Increase HBV Vaccinations in STD Clinics
Brief Title: Interventions to Increase HBV Vaccinations in Sexually Transmitted Disease (STD) Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Gregory Zimet, Professor of Pediatrics & Clinical Psychology, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 0205-04; R01AI049644 (NIH)
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Hepatitis B Virus
Keywords: Attitude to Health; Communication; Intervention Studies; Health Promotion; Psychology, Medical; Sexual Behavior; Behavioral Research; Vaccination
MeSH Terms: conditions — Hepatitis B; Communication; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: 2 X 3 Factorial Design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Non-Framed-Offered (Experimental): Non-Framed, Information Only Condition. Vaccine Offered.
  Interventions: Behavioral: Non-Framed-Offered
- Non-Framed-Recommended (Experimental): Non-Framed, Information Only Condition. Vaccine Recommended.
  Interventions: Behavioral: Non-Framed-Recommended
- Gain-Framed-Offered (Experimental): Gain-Framed Intervention emphasizes the benefits associated with receiving HBV vaccine. Vaccine Offered.
  Interventions: Behavioral: Gain-Framed-Offered
- Gain-Framed-Recommended (Experimental): Gain-Framed Intervention emphasizes the benefits associated with receiving HBV vaccine. Vaccine Recommended.
  Interventions: Behavioral: Gain-Framed-Recommended
- Loss-Framed-Offered (Experimental): Loss-Framed Intervention emphasizes the risks associated with not receiving HBV vaccine. Vaccine Offered.
  Interventions: Behavioral: Loss-Framed-Offered
- Loss-Framed-Recommended (Experimental): Loss-Framed Intervention emphasizes the risks associated with not receiving HBV vaccine. Vaccine Recommended.
  Interventions: Behavioral: Loss-Framed-Recommended

INTERVENTIONS:
Behavioral: Non-Framed-Offered — Subjects received information only and are offered the vaccine.
  Arms: Non-Framed-Offered
Behavioral: Non-Framed-Recommended — Subjects receive information only and are recommended the vaccine.
  Arms: Non-Framed-Recommended
Behavioral: Gain-Framed-Offered — Subjects receive gain-framed messages and are offered the vaccine.
  Arms: Gain-Framed-Offered
Behavioral: Gain-Framed-Recommended — Subjects receive gain-framed messages and are recommended the vaccine.
  Arms: Gain-Framed-Recommended
Behavioral: Loss-Framed-Offered — Subjects receive loss-framed messages and are offered the vaccine.
  Arms: Loss-Framed-Offered
Behavioral: Loss-Framed-Recommended — Subjects receive loss-framed messages and are recommended the vaccine.
  Arms: Loss-Framed-Recommended

SUMMARY:
The goal of this study is to evaluate two sets of interventions to increase acceptance of hepatitis B virus (HBV) vaccination in patients attending sexually transmitted disease (STD) clinics. The 1st set of interventions, with 3 levels, is based on message framing. The 3 levels are: 1. information only; 2. gain-framed message; and 3. loss-framed message. The 2nd set of interventions, with 2 levels, involves how the vaccine is recommended by the health care provider. The 2 levels are: 1. HBV vaccine offered; and 2. HBV vaccine recommended. The outcome of interest is1st dose acceptance.

DETAILED DESCRIPTION:
The goal of this study is to evaluate two sets of interventions to increase acceptance of hepatitis B virus (HBV) vaccination in patients attending sexually transmitted disease (STD) clinics. The 1st specific aim is to assess the effect of message-framing on vaccine acceptance. Framing theory suggests that positively framed messages (i.e., benefits of getting vaccine) are more effective than negatively framed messages (i.e., dangers of not getting vaccine) in stimulating preventive health behaviors. Research on Framing Theory and engagement in health behaviors suggests also that the effects may be moderated by other attitudinal factors, including perceived risk of the behavior and degree of involvement in the message. The 2nd aim is to evaluate the effect of provider-based interventions. Prior research suggests that recommendations by health providers are very important in patients' decisions regarding acceptance of health care procedures. Patients (18 years and older) will be recruited and followed from Chicago and Indianapolis STD clinics during routine medical visits. An audio computer-assisted self-interview (A-CASI) will cover demographics, risk behaviors, and perceived risk associated with vaccination. Subjects then will be randomized to receive a gain-framed, loss-framed, or information only message regarding HBV immunization (also delivered by A-CASI). Upon completion of the message-framing intervention, subjects will complete additional attitude questions via A-CASI. Upon completion of the A-CASI subjects will be randomly assigned to one of two provider intervention conditions: 1. vaccine offered or 2. vaccine recommended. For both conditions free HBV immunization will be provided by a nurse practitioner. Subsequently, postcard reminders will be sent and phone call reminders made for follow-up appointments for those receiving the first and second doses of vaccine. The primary outcome measure is HBV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older males and females
* No prior self-reported history of HBV immunization or infection
* Fluent in English
* Not known to be HIV positive.

Exclusion Criteria:

* Under age 18
* Received any prior HBV vaccination
* Prior infection of Hepatitis B
* Unable to read or comprehend the English language
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1747 (Actual)
Dates: Start 2003-06; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Chicago Department of Public Health, Chicago, Illinois
  - Bell Flower Clinic, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cox AD, Cox D, Zimet G. Promoting prevention and early detection: The impact of message framing, product function and perceived product risk. J Marketing 2006;70:79-91.
- [Derived] Kasting ML, Head KJ, Cox D, Cox AD, Zimet GD. The effects of message framing and healthcare provider recommendation on adult hepatitis B vaccination: A randomized controlled trial. Prev Med. 2019 Oct;127:105798. doi: 10.1016/j.ypmed.2019.105798. Epub 2019 Aug 9. PMID 31404569

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Framed-Offered | Non-Framed-Recommended | Gain-Framed-Offered | Gain-Framed-Recommended | Loss-Framed-Offered | Loss-Framed-Recommended
Started | 299 | 284 | 292 | 288 | 291 | 293
Completed | 299 | 284 | 292 | 288 | 291 | 293
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Framed-Offered | Non-Framed-Recommended | Gain-Framed-Offered | Gain-Framed-Recommended | Loss-Framed-Offered | Loss-Framed-Recommended | Total
Number analyzed (Participants) | 299 | 284 | 292 | 288 | 291 | 293 | 1747
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (9.7) | 31.8 (9.8) | 31.2 (9.8) | 31.7 (9.4) | 32.1 (10.1) | 32.3 (10.6) | 31.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 179 | 175 | 166 | 179 | 177 | 1054
  Male | 121 | 105 | 117 | 122 | 112 | 116 | 693
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 9 | 8 | 6 | 9 | 48
  Not Hispanic or Latino | 284 | 272 | 278 | 275 | 282 | 278 | 1669
  Unknown or Not Reported | 8 | 3 | 5 | 5 | 3 | 6 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 2 | 0 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 252 | 233 | 239 | 233 | 236 | 233 | 1426
  White | 32 | 37 | 37 | 38 | 35 | 45 | 224
  More than one race | 8 | 8 | 5 | 6 | 7 | 9 | 43
  Unknown or Not Reported | 6 | 5 | 9 | 10 | 12 | 4 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 299 | 284 | 292 | 288 | 291 | 293 | 1747

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Doses of HBV Vaccine Received
Description: Mean Number of HBV vaccine doses received over an 8-month period, including the clinic visit. Count values ranged from 0 to 3 doses.
Time Frame: Day of research visit with 8 month follow-up
Measure: Mean (Standard Deviation); unit: Doses of HBV Vaccine
Arm/Group | Non-Framed-Offered | Non-Framed-Recommended | Gain-Framed-Offered | Gain-Framed-Recommended | Loss-Framed-Offered | Loss-Framed-Recommended
Number analyzed (Participants) | 299 | 284 | 292 | 288 | 291 | 293
Doses of HBV Vaccine | .78 (1.00) | .85 (1.02) | .94 (1.11) | .98 (1.06) | .81 (1.04) | 1.10 (1.14)
Statistical Analysis 1: Comparison: Gain-Framed-Offered vs Gain-Framed-Recommended vs Loss-Framed-Offered vs Loss-Framed-Recommended; The two gain-framed groups were compared to the two loss-framed groups using poisson regression; Test type: Superiority; p = .885, Regression, Poisson; Risk Ratio (RR) = 0.99, 95% CI 2-sided [.88 to 1.12]
Statistical Analysis 2: Comparison: Non-Framed-Offered vs Non-Framed-Recommended vs Gain-Framed-Offered vs Gain-Framed-Recommended vs Loss-Framed-Offered vs Loss-Framed-Recommended; Groups receiving any framed interventions (gain-framed or loss-framed) were compared to those in the two non-framed control groups; Test type: Superiority; p < .01, Regression, Poisson; Risk Ratio (RR) = 1.17, 95% CI 2-sided [1.06 to 1.31]
Statistical Analysis 3: Comparison: Non-Framed-Offered vs Non-Framed-Recommended vs Gain-Framed-Offered vs Gain-Framed-Recommended vs Loss-Framed-Offered vs Loss-Framed-Recommended; The 3 vaccine-recommended groups were compared with the 3 vaccine-offered groups using poisson regression; Test type: Superiority; p < .01, Regression, Poisson; Risk Ratio (RR) = 1.16, 95% CI 2-sided [1.05 to 1.28]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Non-Framed-Offered | Non-Framed-Recommended | Gain-Framed-Offered | Gain-Framed-Recommended | Loss-Framed-Offered | Loss-Framed-Recommended
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/284 | 0/292 | 0/288 | 0/291 | 0/293
Serious Adverse Events (participants affected / at risk) | 0/299 | 0/284 | 0/292 | 0/288 | 0/291 | 0/293
Other Adverse Events (participants affected / at risk) | 0/299 | 0/284 | 0/292 | 0/288 | 0/291 | 0/293

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No